CLINICAL TRIAL: NCT05598411
Title: Efficacy of CST1-Guided Oral Glucocorticoid Therapy for Chronic Rhinosinusitis With Polyps
Brief Title: CST1-Guided Oral Glucocorticoids Management for CRSwNP
Acronym: COMPASS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR-COMPASS
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Glucocorticoids
MeSH Terms: interventions — Glucocorticoids; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Glucocorticoids group (Experimental): Intervention Period：oral glucocorticoids（methylprednisolone 24mg qd, 2-week duration）+nasal spray （Budesonide Nasal Spray 64ug per Nostril, bid, 2-week duration） follow-up period：nasal spray（Budesonide Nasal Spray 64ug per Nostril, bid, 24-week duration）
  Interventions: Drug: Oral Glucocorticoids
- Placebo group (Placebo Comparator): Intervention Period：oral placebo+nasal spray（oral placebo 24mg qd, 2-week duration）+nasal spray （Budesonide Nasal Spray 64ug per Nostril, bid, 2-week duration） follow-up period：nasal spray（Budesonide Nasal Spray 64ug per Nostril, bid, 24-week duration）
  Interventions: Drug: Oral placebo

INTERVENTIONS:
Drug: Oral Glucocorticoids — methylprednisolone 24mg qd, 2-week duration
  Other Names: methylprednisolone
  Arms: Oral Glucocorticoids group
Drug: Oral placebo — oral placebo 24mg qd, 2-week duration
  Arms: Placebo group

SUMMARY:
Topical and systemic steroids constitute the first choice in medical treatment for nasal polyps. Glucocorticoids sensitivity is significantly correlated with CST1 in nasal secretions. The goal of this randomized, double-blind, placebo-controlled clinical trial is to clarify the efficacy of a short course of CST1-guided oral glucocorticoids therapy for chronic rhinosinusitis with nasal polyps. Subjects were randomized to receive either oral glucocorticoids or oral placebo for 2 weeks. Endoscopic polyp score, Total Nasal Symptom Score(TNSS), SNOT-22 score, Cystatin 1 and other biomarkers were evaluated before and after the treatment. Researchers will compare oral glucocorticoids group and oral placebo group to test CST1 predictive model of glucocorticoid therapy for Chronic Rhinosinusitis with Polyps.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old；
2. All meet the diagnostic criteria of CRSwNP in EPOS2020;
3. Investigator-assessed endoscopic bilateral Nasal Polyp Size Score (NPSS) was greater than or equal to 4 (minimum score of 2 per nasal cavity);
4. Patients with asthma were in a stable state, with FEV1 > 50% of the predicted value or 50% of the optimal value of personal FEV1; (5) Good compliance, able to complete clinical observation.

Exclusion Criteria:

1. Medication history of oral glucocorticoids within 3 months before enrollment, antibiotics within 2 weeks;
2. Oral glucocorticoid contraindications, such as diabetes, femoral head necrosis, gastric ulcer, etc.;
3. Any nasal and/or sinus surgery within 3 months before enrollment;
4. Patients have conditions or comorbidities that may preclude evaluation of the primary efficacy endpoint, such as: unilateral posterior nasal polyp of maxillary sinus, acute rhinitis, nasal infection or upper respiratory tract at the screening period or within 2 weeks before the screening period infection, acute asthma attack within 4 weeks, current drug-induced rhinitis, allergic fungal sinusitis (AFRS), benign or malignant tumor of nasal cavity；
5. Important clinical comorbidities that may interfere with clinical effectiveness, including but not limited to: active upper or lower respiratory tract infection, cystic fibrosis, eosinophilic granuloma with polyvasculitis (Churg-Strauss syndrome), granulomatosis with polyangiitis (Wegener's granulomatosis), Young's syndrome, etc.;
6. Accompanying serious diseases or recurrent chronic diseases with poor systemic control, such as (but not limited to), active infection, cardiovascular disease, tuberculosis or other pathogen infection, diabetes, autoimmune disease, HIV, hepatitis B, Hepatitis C or parasitic diseases, malignant tumors, etc.;
7. Subjects with severe liver and kidney function injury; such as, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2 times the upper limit of normal, serum creatinine > the upper limit of normal value;
8. Known or suspected immunosuppression, including a history of invasive opportunistic infections (such as tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pulmonary cysts, aspergillosis), even if the infection has subsided;
9. Women who were pregnant or planned to become pregnant during the study, or who were breastfeeding;
10. Subjects who were fertile but were reluctant to use medically approved and effective contraception;
11. Those with a history of alcohol or drug abuse;
12. Those who believed the patient had other medical or non-medical conditions that were not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-17 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The change in endoscopic polyp score | Baseline, week 2, week 6, week 10, week 14, week 18, week 22, week 26
  Bilateral polyp volume size described using the Nasal Polyp Size Score (NPSS) score. (0 - 4 points per side: 0 = no polyp; 1 = small polyp in the middle meatus, not reaching the inferior border of the middle turbinate; 2 = small polyp in the middle meatus, reaching the inferior border of the middle turbinate; 3 = large polyp protruding from the middle meatus, not reaching the inferior border of the inferior turbinate; 4 = large polyp that almost causes most or complete obstruction of the nasal cavity.)

SECONDARY OUTCOMES:
The change in Total Nasal Symptom Score（TNSS） | Baseline, week 2, week 6, week 10, week 14, week 18, week 22, week 26
  Total Nasal Symptom Score was are graded on a 3-point scale. (0= no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms).
The change in SNOT-22 score | Baseline, week 2, week 6, week 10, week 14, week 18, week 22, week 26
  The 22-item Sino-nasal outcome test (SNOT-22) was used to evaluate the changes in symptoms of patients. According to the severity of symptoms caused by RCRS, each item was divided into 6 levels: no distress (0 points), mild distress (1 point), mild distress (2 points) ), moderate distress (3 points), severe distress (4 points), very severe distress (5 points). The higher the score, the more severe the symptoms, and the final total score of the item is counted.
The change in asthma ACQ Score | Baseline, week 2, week 6, week 10, week 14, week 18, week 22, week 26
  For patients with asthma, we assessed the change of asthma symptoms through the Asthma Control Questionnaire(ACQ). Each question was scored on a scale of 0 to 6 according to the severity. The result score of each item was averaged. A score of <0.75 indicated that the asthma had been completely controlled; a score of 0.75-1.5 indicates well-controlled asthma; a score of >1.5 indicates that asthma is not controlled.
The change of CST1 | Baseline, week 2, week 6, week 10, week 14, week 18, week 22, week 26
  The change of Cystatin 1
The change of biomarker | Baseline, week 2, week 6, week 10, week 14, week 18, week 22, week 26
  Changes in expression levels of biomarker in nasal brush exfoliated cells, nasal secretions and nasal microbes.
The change in AE / SAE recording | Baseline, week 2, week 6, week 10, week 14, week 18, week 22, week 26
  Any adverse event
The needs of upgrading treatment | Baseline, week 2, week 6, week 10, week 14, week 18, week 22, week 26
  The needs of upgrading treatment includes surgery, oral glucocorticoids or monoclonal antibodies treatment.
The change of inflammatory cell | Baseline, week 2, week 26
  The change of inflammatory cell in nasal polyps

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Study Chair — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No